CLINICAL TRIAL: NCT00851084
Title: Randomized, Multinational, Study Of Aflibercept And Modified FOLFOX6 As First-Line Treatment In Patients With Metastatic Colorectal Cancer
Brief Title: Study of Aflibercept And Modified FOLFOX6 As First-Line Treatment In Patients With Metastatic Colorectal Cancer
Acronym: AFFIRM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFC10668; EudraCT 2008-004178-41
Record Dates: First submitted 2009-02-24; First posted 2009-02-25 (Estimated); Results first posted 2013-06-25 (Estimated); Last update posted 2016-06-07 (Estimated); Status verified 2016-05

CONDITIONS: Colorectal Neoplasms; Neoplasm Metastasis
Keywords: Angiogenesis; Colon cancer; Rectal cancer; Oxaliplatin
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Colonic Neoplasms; Rectal Neoplasms | interventions — aflibercept; Oxaliplatin; Fluorouracil; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- mFOLFOX6 only (Active Comparator): modified FOLFOX6 chemotherapy regimen
  Interventions: Drug: oxaliplatin; Drug: 5-FU; Drug: Folinic Acid
- mFOLFOX6 + aflibercept (Experimental): modified FOLFOX6 chemotherapy regimen in combination with aflibercept
  Interventions: Drug: aflibercept; Drug: oxaliplatin; Drug: 5-FU; Drug: Folinic Acid

INTERVENTIONS:
Drug: aflibercept — administration: IV infusion
  Other Names: ZALTRAP™; AVE0005
  Arms: mFOLFOX6 + aflibercept
Drug: oxaliplatin — administration: IV infusion
Drug: 5-FU — administration: IV infusion
Drug: Folinic Acid — administration: IV infusion

SUMMARY:
The primary objective of the study is to estimate the progression-free survival rate at 12 months for the two arms of the study.

Secondary objectives include the evaluation of overall objective response rate to treatment, progression-free survival, overall survival, safety and documentation of potential immunogenicity of aflibercept.

This study was a non-comparative randomized trial and was not powered for a comparison of any of the efficacy endpoints.

Rather, the aim of the trial was to get, for all endpoints, an estimation of the efficacy and safety of aflibercept combined with a modified FOLFOX6 regimen. In such type of non-comparative randomized trial, the control FOLFOLX6 arm was intended to only act as a check on the similarity of the current patients to the historical controls with respect to clinical outcome when given FOLFOX6 treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven adenocarcinoma of the colon or the rectum
* Metastatic disease not amenable to potentially curative treatment

Exclusion Criteria:

* Prior therapy for metastatic cancer of the colon or the rectum
* Prior treatment with angiogenesis inhibitors

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Actual)
Dates: Start 2009-02; Primary Completion 2011-04 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Zalcberg, MD, Principal Investigator — Peter Mc Callum Cancer Centre, Melbourne, Australia
Locations (37):
- Australia (3):
  - Sanofi-Aventis Investigational Site Number 036004, Douglas
  - Sanofi-Aventis Investigational Site Number 036001, Hunter Region Mail Centre
  - Sanofi-Aventis Investigational Site Number 036003, Hunter Region Mail Centre
- Germany (7):
  - Sanofi-Aventis Investigational Site Number 276003, Berlin
  - Sanofi-Aventis Investigational Site Number 276007, Dresden
  - Sanofi-Aventis Investigational Site Number 276001, Hanover
  - Sanofi-Aventis Investigational Site Number 276006, Homberg (Efze)
  - Sanofi-Aventis Investigational Site Number 276004, Mannheim
  - Sanofi-Aventis Investigational Site Number 276002, Münster
  - Sanofi-Aventis Investigational Site Number 276005, Recklinghausen
- Italy (5):
  - Sanofi-Aventis Investigational Site Number 380005, Bari
  - Sanofi-Aventis Investigational Site Number 380001, Florence
  - Sanofi-Aventis Investigational Site Number 380002, Milan
  - Sanofi-Aventis Investigational Site Number 380003, Taormina
  - Sanofi-Aventis Investigational Site Number 380004, Torino
- Russia (3):
  - Sanofi-Aventis Investigational Site Number 643002, Pyatigorsk
  - Sanofi-Aventis Investigational Site Number 643005, Saint Petersburg
  - Sanofi-Aventis Investigational Site Number 643001, Sochi
- South Korea (8):
  - Sanofi-Aventis Investigational Site Number 410003, Busan
  - Sanofi-Aventis Investigational Site Number 410004, Cheongju-si
  - Sanofi-Aventis Investigational Site Number 410005, Daegu
  - Sanofi-Aventis Investigational Site Number 410002, Daejeon
  - Sanofi-Aventis Investigational Site Number 410007, Goyang-Si, Gyeonggi-Do
  - Sanofi-Aventis Investigational Site Number 410006, Seoul
  - Sanofi-Aventis Investigational Site Number 410001, Seoul
  - Sanofi-Aventis Investigational Site Number 410008, Ulsan
- Spain (6):
  - Sanofi-Aventis Investigational Site Number 724005, Barcelona
  - Sanofi-Aventis Investigational Site Number 724004, Madrid
  - Sanofi-Aventis Investigational Site Number 724001, Madrid
  - Sanofi-Aventis Investigational Site Number 724002, Sabadell
  - Sanofi-Aventis Investigational Site Number 724007, Santiago de Compostela
  - Sanofi-Aventis Investigational Site Number 724003, Valencia
- United Kingdom (5):
  - Sanofi-Aventis Investigational Site Number 826004, Leeds
  - Sanofi-Aventis Investigational Site Number 826001, Leicester
  - Sanofi-Aventis Investigational Site Number 826002, Manchester
  - Sanofi-Aventis Investigational Site Number 826003, Slough
  - Sanofi-Aventis Investigational Site Number 826005, Southampton

REFERENCES:
- [Result] Folprecht G, Pericay C, Saunders MP, Thomas A, Lopez Lopez R, Roh JK, Chistyakov V, Hohler T, Kim JS, Hofheinz RD, Ackland SP, Swinson D, Kopp M, Udovitsa D, Hall M, Iveson T, Vogel A, Zalcberg JR. Oxaliplatin and 5-FU/folinic acid (modified FOLFOX6) with or without aflibercept in first-line treatment of patients with metastatic colorectal cancer: the AFFIRM study. Ann Oncol. 2016 Jul;27(7):1273-9. doi: 10.1093/annonc/mdw176. Epub 2016 Apr 18. PMID 27091810

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were 268 patients screened (informed consent signed) for this study. Of these screened patients, 236 patients were subsequently randomly assigned to treatments. 32 patients were screen failures.
Groups:
- mFOLFOX6 Only: modified FOLFOX6
- mFOLFOX6 + Aflibercept: modified FOLFOX6 in combination with aflibercept
Period: Overall Study
Arm/Group | mFOLFOX6 Only | mFOLFOX6 + Aflibercept
Started | 117 | 119
Completed | 0 (Participants continued treatment until they met treatment discontinuation criteria.) | 0 (Participants continued treatment until they met treatment discontinuation criteria.)
Not Completed | 117 | 119
Not completed — Randomized but not treated | 1 | 0
Not completed — Adverse Event | 26 | 36
Not completed — Disease progression | 52 | 47
Not completed — Poor compliance to protocol | 1 | 1
Not completed — Physician Decision | 13 | 14
Not completed — Consent withdrawn | 0 | 2
Not completed — Withdrawal by Subject | 11 | 12
Not completed — Metastatic surgery | 6 | 6
Not completed — Other | 7 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | mFOLFOX6 Only | mFOLFOX6 + Aflibercept | Total
Number analyzed (Participants) | 117 | 119 | 236
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.4 (9.7) | 61.8 (9.0) | 62.1 (9.4)
Age, Customized [Number; unit: Participants]
  <65 | 65 | 70 | 135
  >=65 but <75 | 43 | 45 | 88
  >=75 | 9 | 4 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 43 | 92
  Male | 68 | 76 | 144
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian/White | 90 | 97 | 187
  Black | 0 | 1 | 1
  Asian/Oriental | 27 | 20 | 47
  Other | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United Kingdom | 22 | 28 | 50
  Korea, Republic of | 26 | 20 | 46
  Germany | 18 | 24 | 42
  Spain | 24 | 18 | 42
  Russian Federation | 15 | 15 | 30
  Italy | 10 | 5 | 15
  Australia | 2 | 9 | 11
Body Surface Are (BSA) [Mean (Standard Deviation); unit: m^2] | 1.8 (0.2) | 1.8 (0.2) | 1.8 (0.2)

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) Rate at 12 Months
Description: PFS rate at 12 months was defined as the percentage of patients alive without disease progression at 12 months after randomization. The primary efficacy analysis was based on assessment by the Independent Review Committee (IRC). The study was not powered for comparison of PFS rate at 12 months between the two arms (non-comparative, open-label study). Progression was defined using Response Evaluation Criteria In Solid Tumors (RECIST v1.0), as at least a 20 percent increase in the sum of the longest diameter (LD) of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions and/or unequivocal progression of existing non target-lesions.
Time Frame: 12 months
Population: Analyses of PFS rate was performed in the evaluable patient (EP) population as the primary analysis population. Overall, 9 patients from the randomized population were excluded from the EP population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | mFOLFOX6 Only | mFOLFOX6 + Aflibercept
Number analyzed (Participants) | 111 | 116
percentage of participants | 21.2 [12.2 to 30.3] | 25.8 [17.2 to 34.4]

2. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time from the date of randomization to the date of tumor progression or death from any cause, whichever occurred first. PFS was based on tumor assessment by the Independent Review Committee (IRC). PFS was estimated from Kaplan-Meier Curves.
  The study was not powered for comparison of PFS between the two arms (non-comparative, open-label study).
  Progression was defined using Response Evaluation Criteria In Solid Tumors (RECIST v1.0), as at least a 20 percent increase in the sum of the longest diameter (LD) of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions and/or unequivocal progression of existing non target-lesions.
Time Frame: From the date of the first randomization until the study data cut-off date, 14 April 2011 (approximately 26 months)
Population: Evaluable patient (EP) population. A total of 55 patients (32 in the mFOLFOX6 group and 23 in the mFOLFOX6 + aflibercept group) were without an event at the cutoff date for the PFS analysis by IRC.
Measure: Median (95% Confidence Interval); unit: Months
Units Other Than Participants: Events
Arm/Group | mFOLFOX6 Only | mFOLFOX6 + Aflibercept
Number analyzed (Participants) | 111 | 116
Number analyzed (Events) | 79 | 93
Months | 8.77 [7.622 to 9.265] | 8.48 [7.885 to 9.922]

3. Secondary Outcome: Overall Objective Response Rate (ORR)
Description: Summary of overall objective response rate based on tumor assessment by the Independent Review Committee (IRC) as per Response Evaluation Criteria in Solid Tumours (RECIST) criteria. ORR was defined as the proportion of patients with confirmed Complete Response (CR) or confirmed Partial Response (PR) relative to the total number of patients in the analysis population.
  Per RECIST v 1.0 target lesions evaluation and assessed by tumor imaging: Complete Response (CR): Disappearance of all target lesions; Partial Response (PR): >=30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD.
  The study was not powered for comparison of ORR between the two arms (non-comparative, open-label study).
Time Frame: From the date of the first randomization until the study data cut-off date, 14 April 2011 (approximately 26 months)
Population: Evaluable Patient population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | mFOLFOX6 Only | mFOLFOX6 + Aflibercept
Number analyzed (Participants) | 111 | 116
percentage of participants | 45.9 [36.4 to 55.7] | 49.1 [39.7 to 58.6]

4. Secondary Outcome: Overall Survival (OS)
Description: Overall survival was defined as the time from the date of randomization to the date of death due to any cause. In absence of confirmation of death, survival time was censored at the earliest between the last date the patient was known to be alive and the study cutoff date.
  The study was not powered for comparison of OS between the two arms (non-comparative, open-label study).
Time Frame: From the date of the first randomization until the study data cut-off date, 14 April 2011 (approximately 26 months)
Population: Intent-to-treat population (ITT) - all participants who gave informed consent and were randomized. Of the 268 screened participants, 236 were randomly assigned to treatments, whereas 32 participants were screen failures.
Measure: Median (95% Confidence Interval); unit: months
Units Other Than Participants: Events (Death)
Arm/Group | mFOLFOX6 Only | mFOLFOX6 + Aflibercept
Number analyzed (Participants) | 117 | 119
Number analyzed (Events (Death)) | 50 | 51
months | 22.31 [15.57 to NA] — Insufficient number of participants with events. Data have limited maturity and the Kaplan-Meier estimates of median OS are inherently imprecise. | 19.45 [15.64 to NA] — Insufficient number of participants with events. Data have limited maturity and the Kaplan-Meier estimates of median OS are inherently imprecise.

5. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAE)
Description: Summary of treatment-emergent adverse events in the safety population. The National Cancer Institute Common Terminology Criteria for Adverse Event (NCI-CTCAE), version 3.0 was used in this study to grade the severity of AEs.
Time Frame: From the date of the first randomization up to 30 days after the treatment discontinuation or until TEAE was resolved or stabilized
Population: Of the total 235 patients included in the safety population, 116 patients received mFOLFOX6 and 119 patients received mFOLFOX6 + aflibercept. One patient, randomly assigned to the mFOLFOX6 arm did not receive any study treatment and was therefore excluded from the safety analyses.
Measure: Number; unit: participants
Arm/Group | mFOLFOX6 Only | mFOLFOX6 + Aflibercept
Number analyzed (Participants) | 116 | 119
participants
  Treatment Emergent Adverse Event (TEAE) | 115 | 119
  Grade 3-4 TEAE | 87 | 108
  Treatment emergent Serious Adverse Event (SAE) | 32 | 55
  TEAE leading to death | 2 | 8
  Premature treatment discontinuation | NA — Analysis was limited to mFOLFOX6 + aflibercept arm. | 34
  Permanent treatment discontinuation | 26 | 37

6. Secondary Outcome: Immunogenicity of Intravenous (IV) Aflibercept
Description: The antidrug antibody (ADA) assay was evaluated for participants receiving aflibercept.
Time Frame: Any time post baseline and 90 days after the last infusion of aflibercept, according to baseline status
Population: Participants treated with aflibercept and evaluable for antibody assessment.
Measure: Number; unit: participants
Groups:
- Negative or Missing: Negative or missing antidrug antibody (ADA) assay status at Baseline for those participants treated with aflibercept.
- Positive: Positive antidrug antibody (ADA) assay status at Baseline for those participants treated with aflibercept.
Arm/Group | Negative or Missing | Positive
Number analyzed (Participants) | 112 | 3
participants
  ADA Negative post-baseline | 105 | 1
  ADA Positive (drug specific) post-baseline | 7 | 2
  ADA Negative 90 days after last dose | 45 | 1
  ADA Positive 90 days after last dose | 0 | 1

ADVERSE EVENTS:
Description: Of the total 235 patients included in the safety population, 116 patients received mFOLFOX6 and 119 patients received aflibercept+mFOLFOX6. One patient, randomly assigned to the mFOLFOX6 arm did not receive any study treatment and was therefore excluded from the safety analyses.
Arm/Group | mFOLFOX6 Only | mFOLFOX6 + Aflibercept
Serious Adverse Events (participants affected / at risk) | 32/116 | 55/119
Other Adverse Events (participants affected / at risk) | 114/116 | 117/119
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | mFOLFOX6 Only (N=116) | mFOLFOX6 + Aflibercept (N=119)
Urinary tract infection (Infections and infestations) | 0 | 2
Catheter site infection (Infections and infestations) | 3 | 3
Pneumonia (Infections and infestations) | 1 | 4
Cystitis (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 1 | 0
Neutropenic infection (Infections and infestations) | 1 | 0
Abdominal infection (Infections and infestations) | 1 | 0
Gastroenteritis norovirus (Infections and infestations) | 0 | 2
Infectious peritonitis (Infections and infestations) | 0 | 2
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Neutropenic sepsis (Infections and infestations) | 1 | 1
Bacterial infection (Infections and infestations) | 0 | 1
Bronchopneumonia (Infections and infestations) | 0 | 1
Folliculitis (Infections and infestations) | 0 | 1
Fungaemia (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Pneumonia viral (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 0 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 0 | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 2
Drug hypersensitivity (Immune system disorders) | 0 | 3
Adrenal insufficiency (Endocrine disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 1
Convulsion (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 1 | 0
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 | 1
Vision blurred (Eye disorders) | 1 | 0
Retinal detachment (Eye disorders) | 1 | 0
Sinoatrial block (Cardiac disorders) | 0 | 1
Ventricular arrhythmia (Cardiac disorders) | 0 | 1
Subclavian vein thrombosis (Vascular disorders) | 0 | 1
Circulatory collapse (Vascular disorders) | 1 | 0
Hypertensive crisis (Vascular disorders) | 0 | 1
Lymphatic fistula (Vascular disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 3
Stomatitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 2 | 3
Abdominal pain (Gastrointestinal disorders) | 2 | 2
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 4 | 2
Dysphagia (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 0
Colonic obstruction (Gastrointestinal disorders) | 3 | 0
Melaena (Gastrointestinal disorders) | 1 | 1
Anal fistula (Gastrointestinal disorders) | 0 | 1
Ileal perforation (Gastrointestinal disorders) | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 1
Mechanical ileus (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Subileus (Gastrointestinal disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Bile duct obstruction (Hepatobiliary disorders) | 1 | 0
Pyoderma gangrenosum (Skin and subcutaneous tissue disorders) | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 2
Fatigue (General disorders) | 1 | 2
Pyrexia (General disorders) | 3 | 6
Disease progression (General disorders) | 1 | 4
Medical device complication (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 1
Anastomotic leak (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 | 1
Malignant tumour excision (Surgical and medical procedures) | 0 | 1
Tumour excision (Surgical and medical procedures) | 1 | 0
Social stay hospitalisation (Social circumstances) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | mFOLFOX6 Only (N=116) | mFOLFOX6 + Aflibercept (N=119)
Urinary tract infection (Infections and infestations) | 12 | 12
Nasopharyngitis (Infections and infestations) | 8 | 16
Upper respiratory tract infection (Infections and infestations) | 5 | 6
Neutropenia (Blood and lymphatic system disorders) | 64 | 53
Thrombocytopenia (Blood and lymphatic system disorders) | 25 | 14
Anaemia (Blood and lymphatic system disorders) | 11 | 11
Leukopenia (Blood and lymphatic system disorders) | 10 | 11
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 6
Drug hypersensitivity (Immune system disorders) | 6 | 4
Decreased appetite (Metabolism and nutrition disorders) | 37 | 41
Insomnia (Psychiatric disorders) | 3 | 10
Depression (Psychiatric disorders) | 3 | 7
Peripheral sensory neuropathy (Nervous system disorders) | 35 | 23
Headache (Nervous system disorders) | 9 | 39
Neuropathy peripheral (Nervous system disorders) | 24 | 23
Paraesthesia (Nervous system disorders) | 25 | 18
Polyneuropathy (Nervous system disorders) | 16 | 16
Lethargy (Nervous system disorders) | 13 | 14
Dysgeusia (Nervous system disorders) | 16 | 11
Dizziness (Nervous system disorders) | 11 | 12
Dysaesthesia (Nervous system disorders) | 7 | 7
Neurotoxicity (Nervous system disorders) | 6 | 0
Lacrimation increased (Eye disorders) | 3 | 6
Hypertension (Vascular disorders) | 8 | 64
Deep vein thrombosis (Vascular disorders) | 2 | 7
Phlebitis (Vascular disorders) | 0 | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 15 | 34
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 22
Cough (Respiratory, thoracic and mediastinal disorders) | 14 | 12
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3 | 22
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 8
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 6
Nausea (Gastrointestinal disorders) | 62 | 62
Diarrhoea (Gastrointestinal disorders) | 51 | 69
Stomatitis (Gastrointestinal disorders) | 44 | 60
Constipation (Gastrointestinal disorders) | 31 | 37
Vomiting (Gastrointestinal disorders) | 28 | 34
Abdominal pain (Gastrointestinal disorders) | 25 | 21
Dyspepsia (Gastrointestinal disorders) | 12 | 21
Abdominal pain upper (Gastrointestinal disorders) | 14 | 8
Proctalgia (Gastrointestinal disorders) | 3 | 6
Mouth ulceration (Gastrointestinal disorders) | 1 | 6
Alopecia (Skin and subcutaneous tissue disorders) | 15 | 13
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 6 | 20
Rash (Skin and subcutaneous tissue disorders) | 7 | 6
Dry skin (Skin and subcutaneous tissue disorders) | 6 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 5
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 6 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 11 | 9
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 2
Proteinuria (Renal and urinary disorders) | 1 | 28
Fatigue (General disorders) | 30 | 41
Asthenia (General disorders) | 30 | 24
Pyrexia (General disorders) | 18 | 15
Oedema peripheral (General disorders) | 8 | 13
Weight decreased (Investigations) | 6 | 15
Aspartate aminotransferase increased (Investigations) | 6 | 3
Alanine aminotransferase increased (Investigations) | 6 | 2

LIMITATIONS AND CAVEATS:
The overall survival (OS) data are severely limited due to the low number of events (<50%) in both arms, therefore median OS cannot be accurately estimated due to limitations of available data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator shall have the right to independently publish study results from his site after a multicenter publication, or 12 months after the completion of the study by all sites. He must provide the sponsor a copy of any such publication derived from the study for review and comment at least 45 days (20 days for abstracts) in advance of any submission to a journal, and delay publication till the approval of the publication is given in writing by the Sponsor (not to exceed ninety days).